CLINICAL TRIAL: NCT03168945
Title: Quantifying Infectiousness of Undiagnosed Tuberculosis Cases and the Impact of Enhanced Community-based Active Case Finding Strategy Using Novel Diagnostic Tools: A Randomized Controlled Trial
Brief Title: Xpert Active Case-finding Trial 2: Community-based Active Case-finding for Tuberculosis in South Africa
Acronym: XACT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council, South Africa (Other); National Institutes of Health (NIH) (NIH); University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: XACT-2; OISE-16-62105-1 (Other Grant/Funding Number: U.S. Civilian Research and Development Foundation)
Record Dates: First submitted 2016-12-23; First posted 2017-05-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Tuberculosis
Keywords: Active Case Finding
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel diagnostics arm (Active Comparator): The intervention is to screen a sputum specimen collected on a participant with suspected TB in the community at the point-of-contact in a mobile van using an on-site GeneXpert MTB/RIF machine
  Interventions: Other: GeneXpert MTB/RIF
- Routine screening arm (Placebo Comparator): The control arm is to send a sputum specimen collected on a participant with suspected TB at the mobile van for routine smear microscopy at a laboratory
  Interventions: Other: Smear microscopy

INTERVENTIONS:
Other: GeneXpert MTB/RIF — Screening intervention: novel diagnostic for active case finding (GeneXpert MTB/RIF) for TB collected and performed at point-of-contact in a mobile van
  Other Names: GeneXpert Omni
  Arms: Novel diagnostics arm
Other: Smear microscopy — Screening intervention: routine diagnostic test (smear microscopy) for active case finding for TB on sputum collected at point-of-contact in a mobile van but sent to laboratory
  Arms: Routine screening arm

SUMMARY:
TB kills most people with HIV in Africa. TB is out of control. Radically different approaches to deal with the disease is therefor needed. It is known that intensified case finding works in high HIV prevalence environments. However, the poor performance of conventional diagnostics makes the strategy costly and unpalatable for policy makers. If it can be shown that a package of new diagnostic technologies significantly enhances ease and speed of diagnosis, and time to treatment initiation when using intensified case finding, this will usher the way for further studies and policy adjustments to tackle TB. Thus, the work, if found to be useful, could have major policy implications

The purpose of this study will be to determine the diagnostic yield, impact and feasibility of community-based intensified TB case finding using symptom screening, point-of-care TB testing (Xpert Omni), point-of-care HIV testing and CD4 count (Alere PIMA), if HIV-infected, together with a clinic-based diagnostic package (sputum smear microscopy, MGIT sputum culture, and digital chest radiograph). Additionally, the study will assess the infectiousness of previously undiagnosed TB cases in the community using cough aerosol sampling technology (CASS) and will determine the genomic, transcriptomic and lipidomic profile of TB isolates from patients undergoing CASS sampling. The cost-effectiveness of using a novel TB diagnostic platform (Xpert Omni) for intensified case finding compared to conventional methods will also be evaluated.

~6000 people will be screened to enrol 600 participants with suspected TB. It is expected that using the GeneXpert® Omni POC mobile clinic of 2- to 3-person team of healthcare workers in an inexpensive panel van will substantially reduce the time to treatment initiation, and the proportion of individuals initiating and completing TB treatment. Investigators will also review and follow up Household contacts of active TB participants.

As part of the study investigators will also contribute data and specimens to the RePORT consortium (Regional Prospective Observational Research for Tuberculosis), that aims to create a multinational bank with the primary objective of providing specimens and data to RePORT consortia biomarker researchers and their collaborators over the next decade to achieve a better understanding of the prognosis of TB disease; and the pathogenesis of progression from TB exposure to disease.

DETAILED DESCRIPTION:
Background:

TB kills most people with HIV in Africa. TB is out of control. Healthcare professionals therefore need radically different approaches to deal with the disease. It is known that intensified case finding works in high HIV prevalence environments. However, the poor performance of conventional diagnostics makes the strategy costly and unpalatable for policy makers. If it can be shown that a package of new diagnostic technologies significantly enhances ease and speed of diagnosis, and time to treatment initiation when using intensified case finding, then this will usher the way for further studies and policy adjustments to tackle TB. Thus, the work, if found to be useful, could have major policy implications.

Study hypothesis:

Active community-based case finding using a package of diagnostic tools incorporating the new GeneXpert® Omni will detect untreated highly infectious tuberculosis cases (using cough aerosol sampling) and will reduce time to treatment initiation of confirmed TB cases and will increase the proportion of culture-positive TB cases initiating and completing TB treatment, compared to community based screening using a standard intensive-case finding strategy (smear microscopy).

Study design A randomised controlled trial will be used to compare the two diagnostic packages.

In the initial several months of the study, because of delays in procuring the newest locked in version of the Xpert Omni, investigators will use a mobile GeneXpert® 2 module instrument (and not the GeneXpert® Omni) in the intervention arm.

The study staff will undergo separate training on the GeneXpert Omni platform before implementation in the main study. To ensure seamless continuation and minimise bias investigators will conduct a user appraisal and feasibility questionnaire and assessment as done previously in the Xpert RCT.

Study significance

~6000 people will be screened to enrol 600 participants with suspected TB. Investigators expect to show that using the GeneXpert® Omni POC mobile clinic of 2 to 3-person team of healthcare workers in an inexpensive panel van will substantially reduce the time to treatment initiation, and the proportion of individuals initiating and completing TB treatment. At present, 50% of the TB caseload remains undiagnosed in the community and these cases as transmission sentinels that drive the epidemic. GeneXpert® Omni will be a simple and user-friendly approach to intensive case finding compared to a conventional GeneXpert® machine. The data accumulated here will also be used to model the likely impact of this intervention and its cost-effectiveness. These data have substantial implications for active case finding and public health strategy in TB and HIV endemic countries.

Our preliminary studies have indicated that a third of community-diagnosed index cases are smear-positive. Investigators expect that approximately 25% of participants are CASS positive and therefore highly infectious. Investigators will also interrogate the contacts of these index cases. Uniquely, investigators will be able to quantify the duration AND the magnitude of infectiousness of index cases in the community. Thus, investigators will be able to later to model the impact of our intervention on disease burden.

To the investigators' knowledge, the sputum characteristics of index cases who drive transmission in the community have never been comprehensively characterized. Next generation WGS will be used to compare the M.tb isolates obtained from passive case finding clinical cohorts that have already been completed from the same areas. The investigators have the necessary capability to perform WGS and RNAseq as outlined in our preliminary data. Nile red staining have already been performed on about 400 TB sputum samples. It is likely that the investigators will identify specific molecular biomarkers that, in conjunction with cavitation and HIV status, will predict cases who are more likely to transmit disease. This will generate preliminary data for a larger study that will aim to generate a bio-clinical score to identify high transmission risk index cases. The investigators will also determine levels of hetero-resistance and strain variability in isolates from CASS + participants. This will provide insights into strain variability, evolution, and transmission dynamics in the community.

The RePORT consortium The investigators have also been invited to contribute data and specimens to the RePORT consortium (Regional Prospective Observational Research for Tuberculosis), that aims to create a multinational bank with the primary objective of providing specimens and data to RePORT consortia biomarker researchers and their collaborators over the next decade to achieve a better understanding of the prognosis of TB disease; and the pathogenesis of progression from TB exposure to disease.

Methods Study Sites and Population The study will be conducted in Cape Town within high burden developing communities with high HIV prevalence (15-40%) and at their associated primary care TB clinics. This study will be conducted in congregate settings.

Study procedure Each day during the week, a research nurse together with a local community health care worker (CHC) will travel, to the chosen site to perform community based screening. The vehicle will be equipped with portable awning providing shelter, fold up tables, HIV lateral flow testing capability, POC CD4 count estimator (PIMA), a small portable fold-up cubicle for privacy during sputum acquisition, and facilities to securely house and operate the GeneXpert® Omni machine.

The weekly location for the community-based screening will be mapped out so that the entire community is adequately covered during the study period but will be clustered around community congregate settings. Community members will be encouraged to participate using a loudspeaker and vehicle and community-based advertising.

All Participants will be counselled and tested for HIV using a rapid diagnostic kit as per the national guidelines. A positive HIV result will be confirmed by using a second finger-prick test. Incongruent results will be confirmed by an ELISA blood test. TB screening will depend on HIV status as outlined in the inclusion/exclusion criteria. The rationale for including all HIV-positive participants regardless of symptoms is outlined in "Background" above. Sputum will be collected in portable tents.

All participants undergoing screening will have demographic details, 2 mobile numbers documented and tested, and if possible their addresses will be GPS-mapped. The team of research nurse and CHC will aim to screen between 15-20 consenting community members each morning. Participants found to be either HIV-infected or symptomatic for TB will then undergo randomised to either standard diagnostic tools (sputum smear and culture) or a package of novel diagnostic tools (urine LAM strip testing if HIV-infected, sputum MTB/RIF and culture). An SMS randomisation system will be used. A case record form will be completed for all participants undergoing randomisation to document relevant demographics, past medical, occupational and smoking history, TB symptoms and vital signs. Each patient will then be required to give the following samples at baseline:

1) 2 or 3 sputum samples (>1ml each): 2 samples for GeneXpert® Omni MTB/RIF Assay and MTB culture (arm 1) OR

1 sample for fluorescence smear microscopy and MTB culture (arm 2).

1 sample for bio-banking 2) 25μl blood for POC CD4 testing (only if HIV positive) 3) A Urine Sample (15ml) 4) Whole blood for biobanking (10ml)

Participants unable to spontaneously produce sufficient sputum will undergo sputum induction using the standard protocol and infection control. Participants randomized to arm 1 will have the GeneXpert® assay performed in the van.

Chest X-rays will be performed on the following participants:

All participants with active TB confirmed on GeneXpert, Smear or culture. All asymptomatic HIV positive participants. All participants with negative TB microscopy (HIV negative or positive), with ongoing TB symptoms at the 2-month follow-up visit.

X-rays taken on asymptomatic HIV-positive participants will not be used to drive referral to community health centres and/or to advise on empirical treatment, but will be reviewed after the study is concluded to assess the degree of radiological features of TB in an asymptomatic cohort of ambulant HIV-positive participants.

All newly diagnosed TB cases with POC MTB/RIF testing will be giving a letter to commence immediate TB treatment at the nearest DOTs clinic, and participants receiving smear + culture will be contacted telephonically or with home visits and given a letter to commence treatment. TB clinic registers will be visited for all participants commencing anti-TB treatment to determine patient outcomes and ascertain treatment completion status.

Participants with positive diagnostic tests for TB will be recalled for cough aerosol sample testing (CASS), using a sampling system previously validated. Participants are instructed to cough into the CASS as frequently and as strongly as they can for 5 min. They are rested for 5 min before a second 5-min period of coughing. The CASS uses an impactor with agar plates with pores of different sizes to capture droplets in the respirable range. Plates are read at 1 week to detect contaminants, and then at 3 and 6 weeks to count CFU of MTB, which are confirmed by polymerase chain reaction. Culture+ isolates will be biobanked and DNA will be extracted for WGS.

During this CASS-visit (which will take place prior to the initiation of treatment, but will not delay treatment commencement), the investigators will aim to collect the following samples from participants with positive diagnostic tests for TB:

1) 1 or 2 Sputum samples (>1ml each):

1 sample for biobanking

1. additional sample for smear (for participants randomised to the GeneXpert arm). 2) ±35,5ml (±7 teaspoons) of whole blood for the following: Full blood count (3ml) HbA1c (3ml) Genetic analysis (4ml) PAXGene (2,5ml) PBMC (Peripheral Blood Mononuclear Cell) isolation and storage (10ml) IGRA (interferon-Gamma release assay) (3ml) Whole blood for biobanking (10ml) 3) A saliva sample (6ml)

The following will be sent to the Central Bio-repository as part of the RePORT consortium collected at the defined timepoints:

Whole blood (PAXgene RNA) Whole blood (IGRA) Whole blood (genetic analyses) PBMC Plasma Saliva (genetic analyses) Urine Sputum Extracted host RNA Mtb isolate

Household contacts of sputum culture-positive participants will be contacted and offered screening by symptoms, chest X-ray and induced sputum (2 sputum samples for diagnostic testing if symptomatic or HIV positive, and 1 sample for biobanking), regardless of CASS status. This will enable quantification of infectivity and allow for modelling how early detection of TB in the community could potentially affect transmission dynamics.

The following samples will also be collected at baseline, and will be biobanked with the sputum, for future studies of latent TB infection in close contacts of infectious participants: Blood (26ml), Urine (15ml), Saliva (6ml).

Time-to-diagnosis and time-to treatment initiation will be recorded for all newly diagnosed TB cases and these participants will be referred for anti-TB treatment at the clinic. All smear and/or GeneXpert® negative participants with on-going TB symptoms will be reviewed by the attending clinic doctor and investigated in a standardized way.

ELIGIBILITY:
Inclusion criteria for TB suspects

1. Community participant willing to complete community-based symptom screening, urine testing, blood testing for HIV and/or undergo TB diagnostic tests at the local TB clinic.
2. Provision of informed consent.
3. Has documentation of, or willingness to be tested for HIV infection. HIV testing does not need to be repeated if there is written documentation of a confirmed positive test at any time in the past.
4. HIV-negative adults (older than 18 years) with 1 or more of the following:

   * cough ≥ 2 weeks
   * loss of weight
   * Fever
   * night sweats
   * generalized fatigue
   * haemoptysis
   * chest pain
5. Any HIV+ve adult (older than 18 years).
6. Agrees to the collection and storage of blood, urine, saliva, and sputum specimens for use for future research. (The participant may decline collection of specimens for human genetic research and still be eligible for the study.)

To be eligible for the RePORT sample collection aspect of the study, the participant must have either CXR findings consistent with TB, and/or are sputum smear positive by microscopy or by rapid diagnostic test, such as GeneXpert.

Confirmatory Inclusion criteria for RePORT sample collection

a.) Adults must have pulmonary disease confirmed by culture. i. Mtb identified by culture of expectorated or induced sputum. ii. Mtb identified by culture results from respiratory secretions obtained by broncho-alveolar lavage or bronchial wash may not be used to determine study eligibility.

iii. Mtb identified from either liquid or solid culture is acceptable, and may be from either clinical or study-related specimens.

iv. Those who have extra-pulmonary manifestations of TB in addition to pulmonary TB may also be enrolled.

Participants who fail to meet the confirmatory inclusion criteria noted above will be discontinued from the RePORT aspect of the study. However, specimens that were previously collected from the participant may be retained for use as control specimens, and the participants may still continue participation in the XACT-2 study.

Exclusion criteria for TB suspects

1. Inability to provide informed consent (e.g. mentally impaired).
2. Patients self-presenting to the TB clinics.
3. Patients who have completed TB treatment in the last 2 months or received >1 week (daily or intermittent doses) of any drugs with anti-TB activity within 30 days prior to provisional enrolment, including:

   Any drug or combination of drugs typically used in a multidrug anti-TB therapy (isoniazid [INH], rifampicin, pyrazinamide, ethambutol); Any fluoroquinolone (e.g., ofloxacin, ciprofloxacin, levofloxacin, moxifloxacin, nalidixic acid, sparfloxacin, and gatifloxacin); Any other drugs with anti-TB activity (e.g., clofazamine, aminoglycosides [amikacin, kanamycin], or capreomycin).
4. Plans to move from his/her current residence, which would interfere with the participant's ability to complete all study visits (through the 6-Month Post-Treatment Visit).
5. Has an active psychiatric condition, or alcohol or drug dependence that, in the opinion of the site investigator or designee, might interfere with the ability to give true informed consent and to adhere to the study requirements.
6. Is currently imprisoned.

Inclusion criteria for Household contacts (HHC)

1. Adult (> 18 years old) with significant recent exposure (within the past 6 months) to an adult with untreated or inadequately treated pulmonary TB.
2. No clinical signs or symptoms of active TB that include, but are not limited to: persistent cough, haemoptysis, fever, unintended weight loss or failure to thrive (children), fatigue or lethargy, night sweats, pleuritic chest pain, draining lymph node, or other evidence of extra-pulmonary TB. If clinical signs or symptoms of TB are present, CXR and/or sputum culture results must be included in the overall evaluation to rule out active TB.
3. Has signed a written consent or witnessed oral consent in the case of illiteracy, prior to his/her first sample or other study-specific data being collected.
4. Agrees to the collection and storage of blood, urine, saliva and sputum specimens for use for future research. (The participant may decline collection of specimens for human genetic research and still be eligible for the study.)

Exclusion Criteria for Household contacts

1. Plans to move from his/her current residence, which would interfere with the participant's ability to complete all study visits (through the Month 24 Visit).
2. Has an active psychiatric condition, or alcohol or drug dependence that, in the opinion of the site investigator or designee, might interfere with the ability to give true informed consent and to adhere to the study requirements.
3. Is currently imprisoned.

Exclusion from the RePORT aspect of the study (patients may still be included in the XACT II study)

1. Participants enrolled as active TB cases will be discontinued from the study for the following reasons:

   a. More than 1 week of anti-TB therapy was received before the following minimum required baseline laboratory specimens were collected: i. Sputum for culture and Mtb isolate; ii. Sputum for storage; iii. Blood and plasma; and iv. Urine b. The provisional pulmonary TB diagnosis is not confirmed as defined by the protocol (see Confirmatory Inclusion Criteria listed above); c. An HIV test was not completed within the Month 1 Visit window; d. A study outcome occurred: i. Treatment failure (bacteriologic or clinical); ii. TB relapse (bacteriologic or clinical); iii. Emerging resistance; or iv. Completion of the 6-Month Post-Treatment Visit.
2. Household contacts will be discontinued from the study for the following reasons:

   a. A study outcome occurred: i. Active TB develops before the Month 24 Visit; the participant may enroll as an active TB participant if all eligibility criteria are met; or ii. Completion of the Month 24 Visit.
3. Participants will be discontinued from the study for any of the following reasons:

   1. The participant/parent/legal guardian withdraws consent and/or assent;
   2. The participant is lost to follow-up or moves out of the area;
   3. The participant dies;
   4. The participant was inadvertently enrolled;
   5. The investigator determines that further participation would be detrimental to the health or well-being of the participant;
   6. The study is stopped by a funding organization or other government agency; or
4. The study has to stop for other administrative reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The time-to-treatment of culture-positive TB cases initiating TB treatment in each study arm. | Within 2 months of enrollment, up to 24 months
  Time (in days) as determined by difference between enrolment date and date that treatment is commenced in local TB Clinic attendance register.

SECONDARY OUTCOMES:
The proportion of culture-positive TB cases initiating TB treatment in each study arm. | Within 2 months of enrolment, up to 26 months
  Proportion of culture-positive participants initiating treatment as determined by TC Clinic attendance register.
The proportion of culture-positive TB cases completing 6-months of TB treatment in each study arm. | Through study completion, up to 48 months
  Determined by confirming treatment completion (and discharge) by local TB Clinic.
Accuracy of GeneXpert® Omni MTB/RIF at the point-of-care in a mobile unit. | Through study completion, up to 48 months
  Accuracy of lab-based Xpert determined by inter-rater agreement with paired sample analysed using laboratory-based Xpert).
Feasibility of performing GeneXpert® Omni MTB/RIF at the point-of-care in a mobile unit. | Through study completion, up to 48 months
  Number of study days lost to operational problems with machine or van (recorded daily by study team in daily register). Furthermore, user adherence to test protocol, operator knowledge of the testing procedure, and confidence in the test and satisfaction with its ease of use will be tested by two standardised questionnaires employed and validated in our previous study on active case-finding using lab-based Xpert.
User adherence to methodology of GeneXpert® Omni MTB/RIF at the point-of-care in a mobile unit. | Through study completion, up to 48 months
  Confidence in the test and satisfaction with its ease of use will be tested by a standardised questionnaire employed and validated in our previous study on active case-finding using lab-based Xpert.
User acceptance to methodology of GeneXpert® Omni MTB/RIF at the point-of-care in a mobile unit. | Through study completion, up to 48 months
  Measured by standardised questionnaire assessing user adherence to test protocol, employed and validated in our previous study on active case-finding using lab-based Xpert.
Cost per TB case detected between study arms. | Through study completion, up to 48 months
  Cost-effectiveness analysis to be performed at study conclusion.
Cost per TB case successfully completing treatment between study arms. | Through study completion, up to 48 months
  Cost-effectiveness analysis to be performed at study conclusion.
To contribute data and samples as part of the RePORT consortium in order to achieve a better understanding of the prognosis of TB disease and the pathogenesis of progression from TB exposure to disease. | Through study completion, up to 48 months
  Sputum, Blood, Urine and saliva samples will be collected and biobanked for future analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MBChB, PhD, Principal Investigator — Head of Lung Infection and Immunity Unit and Division and Pulmonology
Locations (1):
- University of Cape Town, Cape Town, Western Province, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calligaro GL, Zijenah LS, Peter JG, Theron G, Buser V, McNerney R, Bara W, Bandason T, Govender U, Tomasicchio M, Smith L, Mayosi BM, Dheda K. Effect of new tuberculosis diagnostic technologies on community-based intensified case finding: a multicentre randomised controlled trial. Lancet Infect Dis. 2017 Apr;17(4):441-450. doi: 10.1016/S1473-3099(16)30384-X. Epub 2017 Jan 5. PMID 28063795
- [Derived] Esmail A, Randall P, Oelofse S, Tomasicchio M, Pooran A, Meldau R, Makambwa E, Mottay L, Jaumdally S, Calligaro G, Meier S, de Kock M, Gumbo T, Warren RM, Dheda K. Comparison of two diagnostic intervention packages for community-based active case finding for tuberculosis: an open-label randomized controlled trial. Nat Med. 2023 Apr;29(4):1009-1016. doi: 10.1038/s41591-023-02247-1. Epub 2023 Mar 9. PMID 36894651